CLINICAL TRIAL: NCT00043017
Title: Contrast-Enhanced Breast MRI For Evaluation Of Patients Undergoing Neoadjuvant Treatment For Locally-Advanced Breast Cancer (I-SPY 1/ACRIN 6657)
Brief Title: Magnetic Resonance Imaging in Women Receiving Chemotherapy for Stage III Breast Cancer
Acronym: ACRIN 6657
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: American College of Radiology Imaging Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000069496; ACRIN 6657 (Other: NCI CIP); CALGB-150012
Record Dates: First submitted 2002-08-05; First posted 2003-01-27 (Estimated); Last update posted 2013-10-09 (Estimated); Status verified 2013-10

CONDITIONS: Breast Cancer
Keywords: stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Magnetic Resonance Spectroscopy; Gadolinium DTPA

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MRI/MRS (Experimental): MRI and MRS examinations with standard imaging, with contrast enhancement using an agent (gadopentetate dimeglumine).
  Interventions: Procedure: MRI/MRS; Radiation: gadopentetate dimeglumine

INTERVENTIONS:
Procedure: MRI/MRS — Serial MRI studies evaluated for prognostic properties related to therapeutic response.
  Other Names: magnetic resonance imaging; magnetic resonance spectoscopy
Radiation: gadopentetate dimeglumine — Imaging agent used for contrast enhancement in each of the MRIs.
  Other Names: contrast enhancing agent; MRI contrast; enhanced MRI

SUMMARY:
RATIONALE: Diagnostic procedures such as magnetic resonance imaging (MRI) may help determine the effectiveness of chemotherapy in killing breast cancer and allow doctors to plan more effective treatment.

PURPOSE: Diagnostic trial to study the effectiveness of MRI in monitoring tumor response in women who are receiving chemotherapy for stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Identify surrogate markers of response to neoadjuvant chemotherapy by contrast-enhanced magnetic resonance imaging (MRI) that are predictive of pathologic remissions and survival in women with stage III breast cancer.
* Identify two groups of patients who have statistically different 3-year disease-free survival using MRI measurements of tumor response to neoadjuvant chemotherapy.
* Determine whether MRI measurements of tumor response after the first course of neoadjuvant chemotherapy can predict which of these patients will ultimately have poor clinical response to chemotherapy.
* Compare the accuracy of MRI vs mammography in predicting the extent of residual disease as determined by histopathology in these patients.
* Determine whether initial MRI tumor characteristics (morphologic and vascular patterns) predict pathological response and/or survival in these patients.
* Estimate the conditional probability of response to paclitaxel based on MRI measurements of response to doxorubicin and cyclophosphamide in these patients.

OUTLINE: This is a multicenter study.

Patients receive an injection of gadopentetate dimeglumine and undergo magnetic resonance imaging (MRI) and magnetic resonance spectroscopy of the breast within 4 weeks before beginning neoadjuvant chemotherapy, 20-28 hours or 48-96 hours after the first course of doxorubicin and cyclophosphamide (Type 1 chemotherapy), between Type 1 chemotherapy and paclitaxel chemotherapy regimens (Type 2 chemotherapy) (MRI only) if the patient continues to Type 2 chemotherapy, and 3-4 weeks after final neoadjuvant chemotherapy treatment (1-2 weeks before surgery).

Patients also undergo mammograms and possibly ultrasounds that coincide with the first and last MRI. Core or needle biopsy is performed after the first MRI but before the first course of Type 1 chemotherapy and between Type 1 chemotherapy and Type 2 chemotherapy (if the patient continues to Type 2 chemotherapy).

Patients are followed every 6 months for 7-10 years.

ELIGIBILITY:
ACRIN 6657 eligibility criteria match that of CALGB Correlative Science trial 150007. Patients with histologically-documented tumors per CALGB criteria that are at least 3 cm who choose to undergo neoadjuvant chemotherapy will be eligible to participate in the Correlative Science and Imaging companion trials (CALGB 150007/ACRIN 6657). The therapeutic regimen will consist of AC followed by a taxane for patients enrolled under the original trial protocol, and will consist of a taxane alone (Type 1) or taxane followed by AC (Type 1 followed by Type 2) for patients enrolled as part of the protocol extension.

1. Inclusion Criteria Specific to the ACRIN 6657 MRI Study 1.1 IRB approval/Signed informed consent 1.2 Patients must have a calculated creatinine clearance of > 30 mL/min (modified Cockcroft and Gault formula) based on a serum creatinine level obtained within 28 days of registration in order to participate.

   Creatinine Clearance for Males: ([140-age (years)] X weight (kg)/(serum creatinine X 72) Creatinine Clearance for Females: Creatinine Clearance (male) X 0.85
2. Exclusion Criteria Specific to the ACRIN 6657 MRI Study 2.1 Pregnancy 2.2 Ferromagnetic prostheses

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Actual)
Dates: Start 2002-05; Primary Completion 2005-05 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Disease-free three-year survival | 3 years

SECONDARY OUTCOMES:
Extent of residual disease | 3 years
Change in the maximum dimension of the tumor over time | 3 years
Change in the tumor volume over time | 3 years
Maximum dimension of tumor size measure by MRI, mammography, and pathology | 3 years
MRI volume | 3 years
MRI peak signal enhancement ratio (SER) | 3 years
SER distribution (percent of tumor in highest SER category) | 3 years
Morphological pattern | 3 years
Change in tumor size by clinical exam | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Nola M. Hylton, PhD, Study Chair — University of California, San Francisco
Locations (11):
- United States (11):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Cancer Research Consortium, Rochester, Minnesota
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas

REFERENCES:
- [Background] Carey LA, Oh D, Sawyer L, et al.: Gene expression subtype and p53 mutational status are correlated among neoadjuvantly treated breast cancers in UNC LCCC9819 and I-SPY1 (CALGB 150007/ACRIN 6657). [Abstract] J Clin Oncol 24 (Suppl 18): A-10048, 552s, 2006.
- [Result] Esserman LJ, Berry DA, Cheang MC, Yau C, Perou CM, Carey L, DeMichele A, Gray JW, Conway-Dorsey K, Lenburg ME, Buxton MB, Davis SE, van't Veer LJ, Hudis C, Chin K, Wolf D, Krontiras H, Montgomery L, Tripathy D, Lehman C, Liu MC, Olopade OI, Rugo HS, Carpenter JT, Livasy C, Dressler L, Chhieng D, Singh B, Mies C, Rabban J, Chen YY, Giri D, Au A, Hylton N; I-SPY 1 TRIAL Investigators. Chemotherapy response and recurrence-free survival in neoadjuvant breast cancer depends on biomarker profiles: results from the I-SPY 1 TRIAL (CALGB 150007/150012; ACRIN 6657). Breast Cancer Res Treat. 2012 Apr;132(3):1049-62. doi: 10.1007/s10549-011-1895-2. Epub 2011 Dec 25. PMID 22198468
- [Result] Esserman LJ, Berry DA, DeMichele A, Carey L, Davis SE, Buxton M, Hudis C, Gray JW, Perou C, Yau C, Livasy C, Krontiras H, Montgomery L, Tripathy D, Lehman C, Liu MC, Olopade OI, Rugo HS, Carpenter JT, Dressler L, Chhieng D, Singh B, Mies C, Rabban J, Chen YY, Giri D, van 't Veer L, Hylton N. Pathologic complete response predicts recurrence-free survival more effectively by cancer subset: results from the I-SPY 1 TRIAL--CALGB 150007/150012, ACRIN 6657. J Clin Oncol. 2012 Sep 10;30(26):3242-9. doi: 10.1200/JCO.2011.39.2779. Epub 2012 May 29. PMID 22649152
- [Result] Hylton NM, Blume JD, Bernreuter WK, Pisano ED, Rosen MA, Morris EA, Weatherall PT, Lehman CD, Newstead GM, Polin S, Marques HS, Esserman LJ, Schnall MD; ACRIN 6657 Trial Team and I-SPY 1 TRIAL Investigators. Locally advanced breast cancer: MR imaging for prediction of response to neoadjuvant chemotherapy--results from ACRIN 6657/I-SPY TRIAL. Radiology. 2012 Jun;263(3):663-72. doi: 10.1148/radiol.12110748. PMID 22623692
- [Result] Lin C, Buxton MB, Moore D, Krontiras H, Carey L, DeMichele A, Montgomery L, Tripathy D, Lehman C, Liu M, Olapade O, Yau C, Berry D, Esserman LJ; I-SPY TRIAL Investigators. Locally advanced breast cancers are more likely to present as Interval Cancers: results from the I-SPY 1 TRIAL (CALGB 150007/150012, ACRIN 6657, InterSPORE Trial). Breast Cancer Res Treat. 2012 Apr;132(3):871-9. doi: 10.1007/s10549-011-1670-4. Epub 2011 Jul 28. PMID 21796368
- [Result] Esserman LJ, Perou C, Cheang M, et al.: Breast cancer molecular profiles and tumor response of neoadjuvant doxorubicin and paclitaxel: The I-SPY TRIAL (CALGB 150007/150012, ACRIN 6657). [Abstract] J Clin Oncol 27 (Suppl 15): A-LBA515, 2009.
- [Result] Hylton N, Blume J, Gatsonis C, et al.: MRI tumor volume for predicting response to neoadjuvant chemotherapy in locally advanced breast cancer: findings from ACRIN 6657/CALGB 150007. [Abstract] J Clin Oncol 27 (Suppl 15): A-529, 2009.
- [Result] Lin C, Moore D, DeMichele A, et al.: Detection of locally advanced breast cancer in the I-SPY TRIAL (CALGB 150007/150012, ACRIN 6657) in the interval between routine screening. [Abstract] J Clin Oncol 27 (Suppl 15): A-1503, 2009.
- [Result] Pradhan SM, Carey L, Edmiston S, et al.: P53 mutation and differential response to neoadjuvant chemotherapy in women with locally advanced breast cancer: results from the I-SPY trial (CALGB 150007/1500012 and ACRIN 6657). [Abstract] J Clin Oncol 27 (Suppl 15): A-11099, 2009.
- [Result] Van 't Veer LJ, Das D, DeMichele A, et al.: Neoadjuvant response in the context of a biologically defined low or high risk tumor has a different clinical consequence, the I-SPY trial (CALGB 150007/150012, ACRIN 6657). [Abstract] 32nd Annual San Antonio Breast Cancer Symposium, December 9-13, 2009, San Antonio, Texas. A-2003, 2009.
- [Result] Wolf DM, Das D, Lenburg ME, et al.: From the lab to the clinic: gene-expression profiles that are associated with Mek-inhibitor sensitivity in vitro are coordinately co-expressed in breast cancer biopsy samples from the I-SPY Trial (CALGB 150007/150012, ACRIN 6657). [Abstract] 32nd Annual San Antonio Breast Cancer Symposium, December 9-13, 2009, San Antonio, Texas. A-2042, 2009.
- [Result] Esserman LJ, van't Veer LJ, Perou C, et al.: Biology of breast cancers that present as interval cancers and at young age should inform how we approach early detection and prevention. [Abstract] 31st Annual San Antonio Breast Cancer Symposium, December 10-14, 2008, San Antonio, Texas. A-6034, 2008.
- [Result] Gomez RE, Zakhireh J, Moore D, et al.: Sentinel node biopsy performed in the neoadjuvant setting for breast cancer: results from the I-SPY TRIAL (CALGB 150007/150012 & ACRIN 6657). [Abstract] 31st Annual San Antonio Breast Cancer Symposium, December 10-14, 2008, San Antonio, Texas. A-202, 2008.
- [Result] Hylton NM, Blume JD, Bernreuter WK, et al.: Comparison of MRI endpoints for assessing breast cancer response to neoadjuvant treatment: preliminary findings of the American College of Radiology Imaging Network (ACRIN) trial 6657. [Abstract] 31st Annual San Antonio Breast Cancer Symposium, December 10-14, 2008, San Antonio, Texas. A-6043, 2008.
- [Result] Livasy C, Carey L, DeMichele A, et al.: Influence of anthracycline- and taxane-based neoadjuvant chemotherapy on tumor HER2 protein expression in locally advanced breast cancers: results from the I-SPY TRIAL (CALGB 150007/150012 & ACRIN 6657). [Abstract] 31st Annual San Antonio Breast Cancer Symposium, December 10-14, 2008, San Antonio, Texas. A-703, 2008.
- [Result] Livasy C, Carey L, DeMichele A, et al.: Biomarkers associated with pathologic complete response to neoadjuvant chemotherapy in women with locally advanced breast cancer: results from the I-SPY TRIAL (CALGB 150007/150012 & ACRIN 6657). [Abstract] 31st Annual San Antonio Breast Cancer Symposium, December 10-14, 2008, San Antonio, Texas. A-5102, 2008.